CLINICAL TRIAL: NCT03853304
Title: A Randomized Trial of Quadruple Fortified Salt for Anemia and Birth Defects Prevention in Southern India
Brief Title: Quadruple Fortified Salt Trial in India
Acronym: QFS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Arogyavaram Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 86613
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Anemia; Folate Deficiency; Vitamin B 12 Deficiency
MeSH Terms: conditions — Anemia; Folic Acid Deficiency; Vitamin B 12 Deficiency | interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Intervention Model Description: After confirming eligibility and informed consent/assent, women will be randomly assigned to one of the 4 intervention arms, using a 2 X 2 factorial design:
  1. Quadruple-fortified salt (QFS; i.e., iron, iodine, folic acid, and vitamin B12)
  2. DFS + folic acid
  3. DFS + vitamin B12; and
  4. Double-fortified salt (DFS; i.e., iron and iodine)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All salt formulations will be similar in taste, appearance, and texture. Salt will be packaged in bags labeled with color codes known only to the salt manufacturers and a statistician unaffiliated with the study. A statistician unaffiliated with this study will generate a random number sequence for intervention allocation. Blinding will be maintained until initial data analysis is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Quadruple-Fortified Salt (QFS) (Experimental): Salt fortified with iron, iodine, folic acid, and vitamin B12
  Interventions: Other: + Folic acid; Other: + Vitamin B12; Other: DFS
- DFS + Folic acid (Experimental): Salt fortified with iron, iodine, and folic acid
  Interventions: Other: + Folic acid; Other: DFS
- DFS + Vitamin B12 (Experimental): Salt fortified with iron, iodine, and vitamin B12
  Interventions: Other: + Vitamin B12; Other: DFS
- Double-fortified salt (DFS) (Active Comparator): Salt fortified with iron and iodine
  Interventions: Other: DFS

INTERVENTIONS:
Other: + Folic acid — Salt fortified with folic acid
  Arms: DFS + Folic acid; Quadruple-Fortified Salt (QFS)
Other: + Vitamin B12 — Salt fortified with vitamin B12
  Arms: DFS + Vitamin B12; Quadruple-Fortified Salt (QFS)
Other: DFS — Salt fortified with iron and iodine

SUMMARY:
Women of reproductive age are at an increased risk of anemia and micronutrient deficiencies. Evidence supports the role of periconceptional nutrition in the development of neural tube defects and other pregnancy complications. Vitamin B12 deficiency is a risk factor for neural tube defects and may modify folate biomarkers that predict neural tube defect risk at the population level. There is an interest in mandatory fortification with vitamin B12 and folic acid for anemia and birth defect prevention. However, there are limited population-representative data needed to inform policy and guidelines. This randomized trial will be conducted to evaluate the efficacy of quadruple-fortified salt (QFS; iron, iodine, folic acid, vitamin B12) in 1,000 women and their households in Southern India.

DETAILED DESCRIPTION:
Women of reproductive age are at increased risk for anemia and micronutrient deficiencies, due in part to social structures and increased nutritional requirements across the conceptional period. Anemia is an important public health problem and has been associated with risk of adverse pregnancy outcomes, including maternal and infant mortality, preterm delivery, and low birth weight. Iron deficiency is the leading cause of anemia worldwide, accounting for 20% to half of the anemia cases. Deficiencies in folate and/or vitamin B12 also result in megaloblastic anemia, and inadequate periconceptional folate and vitamin B12 status have been linked to pregnancy complications, including birth defects.

Neural tube defects are among the most common and debilitating birth defects in the United States and globally. Neural tube defects are structural birth defects that arise when the neural folds fail to fuse entirely during early embryogenesis. It is estimated that there are over 260,000 cases of neural tube defects per year globally, ranging from 1 to 80 per 10,000 births, with higher prevalence in low- and middle-income countries. India has one of the highest burdens of neural tube defects in the world, accounting for over one-third of all neural tube defects globally.

The links between maternal folate status and neural tube defect risk in offspring have been well established. In randomized trials, periconceptional folic acid supplementation reduced the risk of neural tube defects by approximately 70%. Fortification of staple foods with folic acid is one of the most efficacious and cost-effective public health interventions and has been linked to decreased neural tube defects in national folic acid fortification programs. Fortification interventions to date have primarily targeted wheat (and maize) flour, which are not primary staples in some settings with the highest burden of neural tube defects, such as Southern India and China.

There is increasing interest in fortification strategies targeting additional staple foods and micronutrient deficiencies in at-risk populations. Emerging evidence suggests that vitamin B12 deficiency is associated with an increased risk of neural tube defects independent of folate status and may modify red blood cell folate concentrations which are used to predict risk of neural tube defects at the population level. In Southern India, the setting of this randomized trial, rice is the primary staple and folic acid fortification is not currently mandatory. Findings from a recently completed population-based pre-intervention biomarker survey in this setting demonstrated a substantial burden of anemia and micronutrient deficiencies of iron, vitamin B12, and folate in women of reproductive age. Together, these findings underscore the potential benefits of developing additional fortification strategies to deliver folic acid and other micronutrients for prevention of anemia and neural tube defects.

Salt fortification is a promising strategy to prevent multiple micronutrient deficiencies, as it is widely consumed, affordable, and has existing production and distribution systems. In India, salt is one of the most widely consumed and fortifiable foods, and double-fortified salt (i.e., with iron and iodine) is included in the national fortification guidelines and social safety net programs in India for prevention of anemia and iron deficiency. Randomized trials demonstrated that double-fortified salt significantly improved serum ferritin or iron deficiency in women of reproductive age and school children. Findings from meta-analyses suggest that double-fortified salt improves hemoglobin concentrations and decreases risk of anemia; however, findings from double-fortified salt trials in India for anemia have been heterogeneous. For example, in a randomized trial of double-fortified salt among Indian female tea pickers by Haas et al., double-fortified salt improved hemoglobin, serum ferritin, total body iron, and soluble transferrin receptor levels, compared with iodized salt without iron, after adjusting for the respective baseline bio- markers. However, the prevalence of anemia (53%) as well as vitamin B12 (37%) and folate (86%) deficiencies remained high at endpoint. These findings highlight the need to develop additional interventions to target other nutritional causes of anemia and multiple micronutrient deficiencies (i.e., vitamin B12 and folate).

Recent technological advances informed the development of a quadruple-fortified salt - i.e., iodine, iron, folic acid, and vitamin B12, which can be adjusted to the level of salt intake in populations. Quadruple-fortified salt has undergone preliminary testing for organoleptic properties and consumer acceptability and is ready for use in randomized efficacy trials in human populations.

The objective of this randomized trial is to evaluate the efficacy of quadruple-fortified salt-i.e., iodine, iron, folic acid, and vitamin B12-on improving 1) hemoglobin, 2) red blood cell folate and serum folate, and 3) vitamin B12 concentrations, among women of reproductive age in Southern India.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 49 years of age
* Healthy
* Not pregnant or lactating
* Plan to reside in the catchment area of our periconceptional surveillance program for at least two years

Exclusion Criteria:

* Severe anemia (Hemoglobin <8.0 g/dL)
* Reported diagnosis of HIV, malaria infection, or active tuberculosis disease
* Malabsorption disorders (i.e., medical conditions that may affect vitamin B12 absorption or metabolism)
* Stage 2 hypertension (SBP≥140 mm Hg or DBP≥90 mm Hg)
* Glycated hemoglobin (HbA1c) ≥6.5%
* Other serious pre-existing medical conditions (e.g., defined as the need for regular medication use), active infections, or acute illnesses
* Previous pregnancy affected by a neural tube defect (i.e., who have had a fetus diagnosed as affected by a neural tube defect or have given birth to a baby with a neural tube defect) (will be referred to OB/GYN for standard of care, including folic acid supplementation, and excluded)
* Planning to become pregnant (or planning to have a child) in the next 12 months (will be referred to OB/GYN for standard of care, including folic acid supplementation, and be excluded)
* Daily micronutrient supplements (i.e., tablets, capsules, dispersible tablets; ≥4 times in the past week)
* Intramuscular or intravenous interventions containing medications or micronutrients (e.g., iron, vitamin B12, folic acid) in the past 3 months

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Concentrations of erythrocyte folate and serum folate | Endpoint (12 months)
  Erythrocyte folate and serum folate concentrations, nmol/L
Concentrations of hemoglobin | Endpoint (12 months)
  Hemoglobin concentrations, g/dL
Concentrations of vitamin B12 | Endpoint (12 months)
  Vitamin B12 concentrations, pmol/L

SECONDARY OUTCOMES:
Folate deficiency and insufficiency | Endpoint (12 months)
  Erythrocyte (RBC) folate <305.0 nmol/L; <748.0 nmol/L
Anemia | Endpoint (12 months)
  Hemoglobin <12.0 g/dL
Vitamin B12 deficiency and insufficiency | Endpoint (12 months)
  Total vitamin B12 <148.0 pmol/L; <221.0 pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Julia L Finkelstein, MPH SM ScD, Principal Investigator — Cornell University
Locations (1):
- Arogyavaram Medical Centre, Madanapalle, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finkelstein JL, Fothergill A, Johnson CB, Guetterman HM, Bose B, Jabbar S, Zhang M, Pfeiffer CM, Qi YP, Rose CE, Williams JL, Bonam W, Crider KS. Anemia and Vitamin B-12 and Folate Status in Women of Reproductive Age in Southern India: Estimating Population-Based Risk of Neural Tube Defects. Curr Dev Nutr. 2021 Apr 26;5(5):nzab069. doi: 10.1093/cdn/nzab069. eCollection 2021 May. PMID 34027296
- [Background] Finkelstein JL, Fothergill A, Johnson CB, Guetterman HM, Bose B, Jabbar S, Zhang M, Pfeiffer CM, Qi YP, Rose CE, Krisher JT, Ruth CJ, Mehta R, Williams JL, Bonam W, Crider KS. Periconceptional surveillance for prevention of anaemia and birth defects in Southern India: protocol for a biomarker survey in women of reproductive age. BMJ Open. 2020 Oct 29;10(10):e038305. doi: 10.1136/bmjopen-2020-038305. PMID 33122315
- [Background] Finkelstein JL, Guetterman HM, Fothergill A, Johnson CB, Qi YP, Jabbar S, Zhang M, Pfeiffer CM, Rose CE, Yeung LF, Williams JL, Krisher JT, Ruth C, Roy Choudhury D, Venkatramanan S, Haas JD, Kuriyan R, Mehta S, Bonam W, Crider KS. A Randomized Trial of Quadruple-Fortified Salt for Anemia and Birth Defects Prevention in Southern India: Protocol Design and Methods. Curr Dev Nutr. 2023 Feb 21;7(3):100052. doi: 10.1016/j.cdnut.2023.100052. eCollection 2023 Mar. PMID 37181934
- [Background] Finkelstein JL, Fothergill A, Guetterman HM, Johnson CB, Bose B, Qi YP, Rose CE, Williams JL, Mehta S, Kuriyan R, Bonam W, Crider KS. Iron status and inflammation in women of reproductive age: A population-based biomarker survey and clinical study. Clin Nutr ESPEN. 2022 Jun;49:483-494. doi: 10.1016/j.clnesp.2022.02.123. Epub 2022 Mar 5. PMID 35623855
- [Derived] Guetterman HM, Rajagopalan K, Fox AM, Johnson CB, Fothergill A, George N, Krisher JT, Haas JD, Mehta S, Williams JL, Crider KS, Finkelstein JL. A Randomized Crossover Trial of Acceptability of Quadruple-Fortified Salt in Women and their Households in Southern India. J Nutr. 2025 Jan;155(1):322-337. doi: 10.1016/j.tjnut.2024.10.037. Epub 2024 Oct 26. PMID 39490799